CLINICAL TRIAL: NCT04525001
Title: MOGGE PAR-A and PAR-P Scores for Prediction of Adverse Outcomes of Placenta Accreta Spectrum: A Multi-center International Validation Study Protocol
Brief Title: MOGGE PAR Scores for Prediction of Outcomes of PAS
Acronym: PAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Middle-East OBGYN Graduate Education Foundation (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, M.B.B.Ch, M.S.c in Gynecology and Obstetrics, Assiut University
Other Study IDs: PAR scores
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Placenta Accreta Spectrum
Keywords: cesarean section; Uterine preservation; MOGGE PAR score; Hysterectomy; Massive hemorrhage
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Placenta accreta spectrum (PAS) is a set of placentation disorders that are associated with trophoblastic invasion through the physiologic decidual-myometrial junction zone. PAS may be associated with massive obstetric hemorrhage, surgical injuries, maternal intensive care unit (ICU) admission, reoperation, and prolonged hospitalization.

This study aims at estimating the validity of "MOGGE placenta accreta risk-antepartum score" or "MOGGE PAR-A score" in predicting potential outcomes once PAS is diagnosed antenatally. In addition, it evaluates the validity of "MOGGE placenta accreta risk-peripartum score" or "MOGGE PAR-P score" in calculating the probability of the same outcomes using baseline features in conjugation with both disease-and surgery-related peripartum variables,thereby,assist designation of the most suitable management. Finally , MOGGE CON-PAS score was created for the subgroup of women who were subject to conservative management to predict probability of uterine preservation success.

DETAILED DESCRIPTION:
Incidence of PAS has significantly increased in concordance with rising trend of cesarean section delivery (CS) among contemporary population.

Although cesarean hysterectomy, without trying to separate placenta (placenta in-situ), is the standard management of PAS, uterine preservation may be routinely offered to women who are concerned about preserving their uteri and may be considered the primary approach in many institutes all over the world.

The "Placenta Accreta Spectrum International Database (PAS-ID)" is an international database that was launched by Middle-East Obstetrics and Gynaecology Graduate Education (MOGGE) Foundation to conduct the current study.

Eligible patients ,with criteria mentioned in following sections, will be counseled on participation by one of the research team. They will be added to study database by an independent investigator(observing investigator) who will collect baseline data and calculate MOGGE PAR-A score using MOGGE PAR score 1.0 software (available at: https://www.mogge-obgyn.com/clinical-studies). The observing investigator will continue to collect clinical data in subsequent visits, through delivery and postpartum visit to calculate MOGGE PAR-P score at the end of follow-up. If patient management involves a uterus preserving procedure, MOGGE CON-PAS score will be calculated as well(it will be available at: https://www.mogge-obgyn.com/clinical-studies). The observing investigator should not be a part of patients'clinical care team, which should be blinded to the calculated scores. data will be collected using an excel spreadsheet designed for this study. Concerned data include patient age, parity, body mass index,smoking, ethnicity, previous gynecologic surgeries, obstetric complications, gestational age at diagnosis and delivery(in weeks), method of diagnosis, administration of antenatal steroids, indication of delivery, pre-delivery and post-delivery hemoglobin (g/dl), operative management, placental site, degree of placental invasion, type of cesarean incision and its relation to the placenta, intra-operative and postoperative complications, intra-operative blood loss in ml, and transfusion of blood products

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with suspected Placenta Accreta Spectrum (PAS),confirmed by clinical and/ or histo-pathological findings.
* They must be planned to deliver in one of centers recruited in this study.

Exclusion Criteria:

* Women who reject participation or whose diagnosis with PAS is eventually excluded based on clinical and/or histo-pathological findings.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study comprises eligible women in 20 centers (anticipated), representing North-America, South-America, Europe, Africa and Asia (all over the world)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Number of women who experience placenta accreta spectrum related massive blood loss | From skin incision to 24 hours postoperative (Total of 24 hours)
  Blood loss > 2500 ml or intra-operative disseminated intravscular coagulopathy (DIC) or transfusion of 10 or more packed red blood cell units
Number of mothers admitted to intensive care unit | From skin incision to 24 hours postoperative (Total of 24 hours)
  Admission to intensive care unit after delivery
Days of maternal hospitalization after delivery | From Cesarean delivery till hospital discharge (Assessment up to 6 weeks)
  Maternal admission to hospital for more than 7 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Shazly, M.Sc, Principal Investigator — Assiut University

REFERENCES:
- [Background] Jauniaux E, Collins S, Burton GJ. Placenta accreta spectrum: pathophysiology and evidence-based anatomy for prenatal ultrasound imaging. Am J Obstet Gynecol. 2018 Jan;218(1):75-87. doi: 10.1016/j.ajog.2017.05.067. Epub 2017 Jun 24. PMID 28599899
- [Background] Silver RM, Branch DW. Placenta Accreta Spectrum. N Engl J Med. 2018 Apr 19;378(16):1529-1536. doi: 10.1056/NEJMcp1709324. No abstract available. PMID 29669225
- [Background] Society of Gynecologic Oncology; American College of Obstetricians and Gynecologists and the Society for Maternal-Fetal Medicine; Cahill AG, Beigi R, Heine RP, Silver RM, Wax JR. Placenta Accreta Spectrum. Am J Obstet Gynecol. 2018 Dec;219(6):B2-B16. doi: 10.1016/j.ajog.2018.09.042. PMID 30471891
- [Background] Cal M, Ayres-de-Campos D, Jauniaux E. International survey of practices used in the diagnosis and management of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2018 Mar;140(3):307-311. doi: 10.1002/ijgo.12391. Epub 2017 Dec 22. PMID 29149470
- [Background] Shazly SA, Hortu I, Shih JC, Melekoglu R, Fan S, Ahmed FUA, Karaman E, Fatkullin I, Pinto PV, Irianti S, Tochie JN, Abdelbadie AS, Ergenoglu AM, Yeniel AO, Sagol S, Itil IM, Kang J, Huang KY, Yilmaz E, Liang Y, Aziz H, Akhter T, Ambreen A, Ates C, Karaman Y, Khasanov A, Larisa F, Akhmadeev N, Vatanina A, Machado AP, Montenegro N, Effendi JS, Suardi D, Pramatirta AY, Aziz MA, Siddiq A, Ofakem I, Dohbit JS, Fahmy MS, Anan MA; and Middle East Obstetrics and Gynecology Graduate Education (MOGGE) foundation - Artificial intelligence (AI) unit. Prediction of clinical outcomes in women with placenta accreta spectrum using machine learning models: an international multicenter study. J Matern Fetal Neonatal Med. 2022 Dec;35(25):6644-6653. doi: 10.1080/14767058.2021.1918670. Epub 2021 Jul 7. PMID 34233555
- [Background] Mohri M, Rostamizadeh A, Talwalkar A: Foundations of machine learning: MIT press; 2018.
- [Derived] Shazly SA, Anan MA, Makukhina TB, Melekoglu R, Ahmed FUA, Pinto PV, Takahashi H, Ahmed NB, Sayed EG, Elassall GM, Said AE, Fahmy MS, Dawyee DM, Penzhoyan GA, Amirkhanyan AM, Yilmaz E, Celik NZ, Aziz H, Akhter T, Ambreen A, Abdelbadie AS. Placenta accreta risk-antepartum score in predicting clinical outcomes of placenta accreta spectrum: A multicenter validation study. Int J Gynaecol Obstet. 2022 Aug;158(2):424-431. doi: 10.1002/ijgo.13993. Epub 2021 Nov 14. PMID 34674270